CLINICAL TRIAL: NCT02591147
Title: Effectiveness of Silver Diamine Fluoride in Arresting Early Approximal Carious Lesion Progression: A Pilot Study
Brief Title: Silver Diamine Fluoride Pilot Study (SDF)
Acronym: SDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Justine Kolker (Other)
Responsible Party: Sponsor-Investigator, Justine Kolker, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 201509831
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Silver Diamine Fluoride 38% (Active Comparator): Group 1 (SDF 38%) will receive the application of silver diammine fluoride (38% SDF solution) in addition to 5% sodium fluoride varnish to each approximal carious lesion (scores RA1,RA2,RA3) in a posterior tooth (premolar or molar) that is in contact with an adjacent tooth, using super floss, for a duration of 3 minutes under rubber dam isolation.
  Interventions: Device: Silver Diamine Fluoride 38%
- Placebo (Sterile water) (Placebo Comparator): Group 2 Placebo (control) will receive the application of sterile water (placebo) in addition to 5% sodium fluoride varnish to each approximal carious lesion (scores RA1,RA2,RA3) in a posterior tooth (premolar or molar) that is in contact with an adjacent tooth, using super floss, for a duration of 3 minutes under rubber dam isolation.
  Interventions: Device: Group 2 (Placebo)

INTERVENTIONS:
Device: Silver Diamine Fluoride 38% — Group 1 (SDF group) subjects will receive the application of silver diamine fluoride (38% SDF solution) in addition to 5% Fluoride varnish to each approximal incipiency, using super floss, for a duration of 3 minutes under rubber dam isolation.
  Other Names: 38% SDF
  Arms: Silver Diamine Fluoride 38%
Device: Group 2 (Placebo) — Group 2 (Placebo) subjects will receive application of sterile water (placebo) in addition to 5% Fluoride varnish to each approximal incipiency, using super floss, for a duration of 3 minutes under rubber dam isolation.
  Other Names: Sterile Water
  Arms: Placebo (Sterile water)

SUMMARY:
This pilot trial is randomized, double-blind, and placebo-controlled trial with two parallel arms: an intervention group using silver diamine fluoride (SDF) and a placebo group (control). 60 eligible healthy adults will be enrolled in the study and randomly assigned to one of the two treatment groups. Both groups will receive the traditional preventive measures including cleanings, Fluoride varnish, diet analysis and counseling. Study participants will be followed for one year and caries progression will be radiographically monitored.

DETAILED DESCRIPTION:
This pilot study will compare 1) Silver diamine fluoride (SDF) and fluoride varnish to 2) Placebo and fluoride varnish (conventional prevention) in the management of early approximal carious lesions. Early approximal carious lesions refers to decay between teeth, diagnosed with radiographs, not extending more than 1/3 of the way into dentin. Management of early approximal carious lesions refers to halting lesion progression, or encouraging lesion reversal after an early carious lesion is detected.

SDF provides a novel, low-cost intervention option for managing early carious lesions that could potentially bridge the 'gap' between non-operative and operative options; thus, postponing the first placement of a restoration. SDF has been used in arresting carious lesions for more than 100 years. However, SDF has never been tested in the arrest of approximal caries lesions in permanent teeth.

SDF acts to both prevent and arrest tooth decay in multiple ways: 1) it acts on the body of carious lesions by precipitating silver ion into the lesion, thus blocking diffusion pathways for cariogenic acids; 2) it interacts with dental enamel leading to the formation of fluoroapatite crystals making the tooth surface more acid resistant; and 3) the precipitated silver from SDF acts as a bactericidal agent disturbing the formation of cariogenic biofilm.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one approximal caries lesion (scores RA1, RA2, RA3 according to the ICCMS radiographic scoring system) in one of the posterior teeth (premolars and molars) presented with full contact with the adjacent tooth.
* All the surfaces eligible for this study will be included.

Exclusion Criteria:

* The approximal lesion detected in the radiograph has advanced dentine lesion (RB4, RC5, or RC6)
* or is adjacent to a lesion that is either filled or will receive a filling at the time of enrollment.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kanellis, DDS, MS, Principal Investigator — University of Iowa; Justine Kolker, DDS, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenblatt A, Stamford TC, Niederman R. Silver diamine fluoride: a caries "silver-fluoride bullet". J Dent Res. 2009 Feb;88(2):116-25. doi: 10.1177/0022034508329406. PMID 19278981
- [Background] Santos VE Jr, Vasconcelos Filho A, Targino AG, Flores MA, Galembeck A, Caldas AF Jr, Rosenblatt A. A new "silver-bullet" to treat caries in children--nano silver fluoride: a randomised clinical trial. J Dent. 2014 Aug;42(8):945-51. doi: 10.1016/j.jdent.2014.05.017. Epub 2014 Jun 12. PMID 24930870
- [Background] Peng JJ, Botelho MG, Matinlinna JP. Silver compounds used in dentistry for caries management: a review. J Dent. 2012 Jul;40(7):531-41. doi: 10.1016/j.jdent.2012.03.009. Epub 2012 Apr 3. PMID 22484380
- [Background] Mattos-Silveira J, Floriano I, Ferreira FR, Vigano ME, Frizzo MA, Reyes A, Novaes TF, Moriyama CM, Raggio DP, Imparato JC, Mendes FM, Braga MM. New proposal of silver diamine fluoride use in arresting approximal caries: study protocol for a randomized controlled trial. Trials. 2014 Nov 19;15:448. doi: 10.1186/1745-6215-15-448. PMID 25409545
- [Background] Tellez M, Gomez J, Kaur S, Pretty IA, Ellwood R, Ismail AI. Non-surgical management methods of noncavitated carious lesions. Community Dent Oral Epidemiol. 2013 Feb;41(1):79-96. doi: 10.1111/cdoe.12028. PMID 23253076
- [Background] Llodra JC, Rodriguez A, Ferrer B, Menardia V, Ramos T, Morato M. Efficacy of silver diamine fluoride for caries reduction in primary teeth and first permanent molars of schoolchildren: 36-month clinical trial. J Dent Res. 2005 Aug;84(8):721-4. doi: 10.1177/154405910508400807. PMID 16040729
- [Background] Ekstrand KR, Bruun G, Bruun M. Plaque and gingival status as indicators for caries progression on approximal surfaces. Caries Res. 1998;32(1):41-5. doi: 10.1159/000016428. PMID 9438570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silver Diamine Fluoride 38% | Placebo (Sterile Water)
Started | 20 | 21
Completed | 18 | 16
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver Diamine Fluoride 38% | Placebo (Sterile Water) | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Radiographic Change in Dental Cavity
Description: Determine if there is a change in the size of the dental cavity from baseline to 12 months after blinded treatment with either Silver Diamine Fluoride 38% or placebo (sterile water). This measurement will be assessed using radiographic examination to determine if there is either evidence of no radiographic change, radiographic progression, or radiographic regression.
Time Frame: Baseline, 12 months after blinded treatment with either Silver Diamine Fluoride 38% or placebo (sterile water)
Measure: Count of Participants; unit: Participants
Arm/Group | Silver Diamine Fluoride 38% | Placebo (Sterile Water)
Number analyzed (Participants) | 18 | 16
Participants
  No radiographic change | 9 | 11
  Radiographic progression | 3 | 2
  Radiographic regression | 6 | 3

ADVERSE EVENTS:
Time Frame: 1 year from baseline
Arm/Group | Silver Diamine Fluoride 38% | Placebo (Sterile Water)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT02591147/Prot_SAP_000.pdf